CLINICAL TRIAL: NCT03758755
Title: The Effect of Blood Flow Restriction Therapy Following Anterior Cruciate Ligament Reconstruction
Brief Title: Blood Flow Restriction Following ACL Reconstruction
Acronym: BFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Principal Investigator, Edward Chang, MD, Orthopedic Surgeon, Inova Health Care Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-3150
Record Dates: First submitted 2018-11-14; First posted 2018-11-29 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: BFR; ACL; rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BFR Therapy (Experimental): This group will undergo physical therapy exercises per the standard of care, with the addition of Blood Flow Restriction (BFR) utilizing a wide pressure cuff. BFR exercises will be initiated two weeks post-op, and continued for 16 weeks.
  Interventions: Device: Blood Flow Restriction Therapy; Other: ACL Reconstruction rehabilitation
- No BFR (Active Comparator): This group of patients will undergo physical therapy exercises per the current standard of care after their ACL reconstruction without BFR
  Interventions: Other: ACL Reconstruction rehabilitation

INTERVENTIONS:
Device: Blood Flow Restriction Therapy — A wide pressure cuff will be applied to the upper thigh prior to starting strengthening exercises. The cuff is inflated to 80% of resting systolic blood pressure. The cuff remains inflated for the entirety of the exercise (4 sets of a specific movement). Once the exercises are completed, it is deflated for a minimum of one minute before the next type of exercises are started.
  Arms: BFR Therapy
Other: ACL Reconstruction rehabilitation — post-operative rehabilitation according to current standards of care

SUMMARY:
The main objective is to determine the impact of Blood Flow Restriction (BFR) therapy, in comparison to a standard rehabilitation protocol, on preventing atrophy, improving quadriceps strength and improving functional outcomes of patients recovering from ACL reconstruction. The investigators hypothesize that patients undergoing BFR therapy after ACL reconstruction surgery will have better functional outcomes than those undergoing normal rehabilitation without BFR therapy.

DETAILED DESCRIPTION:
Recovery from anterior cruciate ligament (ACL) reconstruction involves early physical therapy to promote muscular development. Traditional training regimens are based on the concept that muscle growth is induced with high resistance exercises of at least 65-70% of 1-repetition maximum. Achieving a high resistance level can be challenging in the early post-surgical patient who may be limited by pain, muscle atrophy, diminished proprioception, and psychological factors. Increasing evidence has suggested that Blood Flow Restriction (BFR) in resistance training, while transmitting a decreased load (25-50% of 1-repetition maximum) across the surgical site, may provide an additional benefit of inducing muscular development similar to that of high intensity exercises .

Augmenting exercises with BFR involves an external pressure cuff applied to the proximal portion of the extremity, which is inflated to a pressure that restricts venous outflow while allowing arterial inflow to continue. This creates a physiologic environment for the patient to gain the hypertrophic effect of high resistance training, though at a lower and safer intensity. Studies suggest that BFR stimulates muscular development through an increase in metabolic stress, muscle fiber recruitment, cell swelling, and protein synthesis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 13-35 years at the time of surgery
2. Anterior Cruciate Ligament (ACL) reconstruction
3. Using a physical therapy center with Blood Flow Restriction capabilities.

Exclusion Criteria:

1. Concomitant ligament reconstruction
2. Concurrent procedures that require delayed weight bearing (ie: High Tibial Osteotomy (HTO), multi-ligament reconstruction, microfracture, etc)
3. History of Deep Vein Thrombosis (DVT)/Pulmonary Embolism (PE)
4. Immunocompromising conditions (ie: Rheumatoid arthritis, chronic steroid use, etc.)
5. History of coagulation disorders or current use of anticoagulants
6. Completion of physical therapy at a location not affiliated with the study
7. Pregnancy

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Chang, MD, Principal Investigator — Orthopedic Surgeon
Locations (1):
- Inova Health System, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hughes L, Paton B, Rosenblatt B, Gissane C, Patterson SD. Blood flow restriction training in clinical musculoskeletal rehabilitation: a systematic review and meta-analysis. Br J Sports Med. 2017 Jul;51(13):1003-1011. doi: 10.1136/bjsports-2016-097071. Epub 2017 Mar 4. PMID 28259850
- [Background] Iversen E, Rostad V, Larmo A. Intermittent blood flow restriction does not reduce atrophy following anterior cruciate ligament reconstruction. J Sport Health Sci. 2016 Mar;5(1):115-118. doi: 10.1016/j.jshs.2014.12.005. Epub 2015 Apr 18. PMID 30356481
- [Background] Ohta H, Kurosawa H, Ikeda H, Iwase Y, Satou N, Nakamura S. Low-load resistance muscular training with moderate restriction of blood flow after anterior cruciate ligament reconstruction. Acta Orthop Scand. 2003 Feb;74(1):62-8. doi: 10.1080/00016470310013680. PMID 12635796
- [Background] Scott BR, Loenneke JP, Slattery KM, Dascombe BJ. Blood flow restricted exercise for athletes: A review of available evidence. J Sci Med Sport. 2016 May;19(5):360-7. doi: 10.1016/j.jsams.2015.04.014. Epub 2015 May 9. PMID 26118847
- [Background] Suga T, Okita K, Takada S, Omokawa M, Kadoguchi T, Yokota T, Hirabayashi K, Takahashi M, Morita N, Horiuchi M, Kinugawa S, Tsutsui H. Effect of multiple set on intramuscular metabolic stress during low-intensity resistance exercise with blood flow restriction. Eur J Appl Physiol. 2012 Nov;112(11):3915-20. doi: 10.1007/s00421-012-2377-x. Epub 2012 Mar 14. PMID 22415101
- [Background] Takada S, Okita K, Suga T, Omokawa M, Morita N, Horiuchi M, Kadoguchi T, Takahashi M, Hirabayashi K, Yokota T, Kinugawa S, Tsutsui H. Blood flow restriction exercise in sprinters and endurance runners. Med Sci Sports Exerc. 2012 Mar;44(3):413-9. doi: 10.1249/MSS.0b013e31822f39b3. PMID 21795999
- [Background] Takarada Y, Takazawa H, Sato Y, Takebayashi S, Tanaka Y, Ishii N. Effects of resistance exercise combined with moderate vascular occlusion on muscular function in humans. J Appl Physiol (1985). 2000 Jun;88(6):2097-106. doi: 10.1152/jappl.2000.88.6.2097. PMID 10846023
- [Background] Yasuda T, Brechue WF, Fujita T, Shirakawa J, Sato Y, Abe T. Muscle activation during low-intensity muscle contractions with restricted blood flow. J Sports Sci. 2009 Mar;27(5):479-89. doi: 10.1080/02640410802626567. PMID 19253083

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from two fellowship trained sports medicine orthopedic surgeons at a large health system from November 2018 to November 2021.
Pre-assignment Details: Of 49 enrolled patients, 45 met inclusion/exclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | BFR Therapy | No BFR
Started | 25 | 20
Completed | 25 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BFR Therapy | No BFR | Total
Number analyzed (Participants) | 25 | 20 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.4 (10.08) | 29.0 (9.41) | 26.8 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 19 | 13 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Laterality [Count of Participants; unit: Participants]
  Right | 16 | 10 | 26
  Left | 9 | 10 | 19
Type of Anterior Cruciate Ligament (ACL) Graft [Count of Participants; unit: Participants] — Graft choices for ACL Reconstruction varied based on surgeon and patient preference, and consisted of Allograft, Bone-Patellar Tendon-Bone Autograft, Hamstring Tendon Autograft, and Quadriceps Tendon Autograft.
  Participants
    Allograft | 2 | 1 | 3
    Bone-Patellar Tendon-Bone Autograft | 15 | 11 | 26
    Hamstring Tendon Autograft | 5 | 5 | 10
    Quadriceps Tendon Autograft | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: International Knee Documentation Committee (IKDC) Questionnaire Score
Description: The International Knee Documentation Committee (IKDC Questionnaire) is a knee-specific patient-reported outcome measure. The IKDC Questionnaire is a subjective scale that provides patients with an overall function score. The questionnaire looks at 3 categories: symptoms, sports activity, and knee function. Scores are obtained by summing the individual items, then transforming the crude total to a scaled number that ranges from 0 to 100. This final number is interpreted as a measure of function with higher scores representing higher levels of function.
Time Frame: Measured preoperatively and at 12 weeks post-op.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | BFR Therapy | No BFR
Number analyzed (Participants) | 25 | 20
score on a scale
  Preoperative visit | 47.40 (8.00) | 50.80 (4.01)
  12 weeks post-op | 61.83 (2.93) | 52.86 (3.25)
Statistical Analysis 1: Comparison: BFR Therapy vs No BFR; Null hypothesis: there is no difference between groups in IKDC score at 12 weeks post-op; Test type: Equivalence — The a priori threshold for statistical significance was set at 0.05; p = 0.0219, t-test, 1 sided

2. Primary Outcome: Visual Analog Score
Description: The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain," with "no pain" corresponding to a VAS score of 0 and "worst pain" corresponding to a VAS score of 10.
Time Frame: Measured preoperatively, at 2-weeks post-op, 6 weeks post-op, and 12 weeks post-op
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | BFR Therapy | No BFR
Number analyzed (Participants) | 25 | 20
score on a scale
  Preoperative visit | 2.36 (0.50) | 3.18 (1.02)
  2 weeks post-op | 2.72 (0.65) | 3.16 (0.63)
  6 weeks post-op | 1.00 (0.26) | 1.51 (0.56)
  12 weeks post-op | 0.29 (0.30) | 1.16 (0.37)
Statistical Analysis 1: Comparison: BFR Therapy vs No BFR; Null hypothesis: there is no difference between groups in VAS score at 12 weeks post-op; Test type: Equivalence — The a priori threshold for statistical significance was set at 0.05; p = 0.008, t-test, 1 sided

3. Primary Outcome: Quadriceps Tendon Strength
Description: We will measure quadriceps tendon strength (closed chain) strength using a hand-held dynamometer placed just distal to the knee joint on the posterior calf with the patient in the supine position. The outcome will be reported biweekly as a percentage of the strength of the contralateral side, and then finally reported as a change in strength from the first measurement to the final measurement. The results reported in this data table refer to the percent strength of the operated leg when compared to the contralateral side. The change in strength results can be found in the statistical analysis section.
Time Frame: Tracked from initiation of therapy 2 weeks post-op through 12 weeks post-op.
Measure: Mean (Standard Error); unit: percent difference to contralateral side
Arm/Group | BFR Therapy | No BFR
Number analyzed (Participants) | 25 | 20
percent difference to contralateral side
  Week 2 | 58.88 (4.45) | 51.35 (5.85)
  Week 4 | 63.68 (3.37) | 66.13 (3.43)
  Week 6 | 75.73 (4.11) | 68.51 (3.33)
  Week 8 | 79.39 (2.07) | 72.88 (3.16)
  Week 10 | 80.22 (2.89) | 78.41 (5.11)
  Week 12 | 85.47 (3.84) | 73.03 (5.31)
Statistical Analysis 1: Comparison: BFR Therapy vs No BFR; This analysis compares the change over time in quadriceps tendon strength between the BFR Therapy group and the No BFR Group. Underlying data was collected on a biweekly basis as the percent difference of the operated knee compared to the contralateral side. This statistical test utilized the null hypothesis that there would be no difference between groups in the change in quadriceps tendon strength over time; Test type: Equivalence — The a priori threshold for statistical significance was set at 0.05; p = 0.011, t-test, 1 sided

4. Primary Outcome: Thigh Circumference
Description: A tape measure will be used to measure the thigh circumference 15 cm proximal to the superior pole of the patella. The outcome will be reported biweekly as a percentage of the contralateral side, and then finally reported as a change in circumference from the first measurement to the final measurement. The results reported in this data table refer to the percent circumference of the operated leg when compared to the contralateral side. The change in circumference results can be found in the statistical analysis section.
Time Frame: Tracked in the perioperative week and then from initiation of therapy 2 weeks post-op through 12 weeks post-op.
Measure: Mean (Standard Error); unit: percent difference to contralateral side
Arm/Group | BFR Therapy | No BFR
Number analyzed (Participants) | 25 | 20
percent difference to contralateral side
  Perioperative | 99.23 (1.65) | 101.62 (2.09)
  2 weeks post-op | 97.02 (1.11) | 97.68 (1.05)
  4 weeks post-op | 94.55 (0.82) | 97.11 (0.94)
  6 weeks post-op | 95.33 (1.05) | 95.55 (0.91)
  8 weeks post-op | 96.03 (0.71) | 95.76 (1.09)
  10 weeks post-op | 96.00 (0.71) | 96.46 (0.90)
  12 weeks post-op | 98.28 (0.61) | 98.27 (0.83)
Statistical Analysis 1: Comparison: BFR Therapy vs No BFR; This analysis compares the change over time in thigh circumference between the BFR Therapy group and the No BFR Group. Underlying data was collected on a biweekly basis as the percent difference of the operated knee compared to the contralateral side. This statistical test utilized the null hypothesis that there would be no difference between groups in the change in thigh circumference over time; Test type: Equivalence — The a priori threshold for statistical significance was set at 0.05; p = 0.223, t-test, 1 sided

5. Primary Outcome: Degrees of Knee Flexion
Description: Degrees of knee flexion will be measured on the operative side by a licensed physical therapist. The outcome will be reported biweekly and then finally reported as a change in degrees from the first measurement to the final measurement. The results reported in this data table refer to the degrees of knee flexion at each reported time point. The change in knee flexion results can be found in the statistical analysis section.
Time Frame: Tracked in the perioperative week and then from initiation of therapy 2 weeks post-op through 12 weeks post-op.
Measure: Mean (Standard Error); unit: degrees
Arm/Group | BFR Therapy | No BFR
Number analyzed (Participants) | 25 | 20
degrees
  Perioperative Week | 51.54 (4.43) | 41.9 (4.22)
  2 weeks post-op | 76.4 (3.53) | 70.00 (5.35)
  4 weeks post-op | 102.02 (3.07) | 91.75 (4.18)
  6 weeks post-op | 121.08 (2.73) | 112.74 (3.74)
  8 weeks post-op | 130.78 (2.74) | 126.22 (3.34)
  10 weeks post-op | 135.35 (2.19) | 130.12 (2.52)
  12 weeks post-op | 137.18 (2.20) | 130.50 (2.59)
Statistical Analysis 1: Comparison: BFR Therapy vs No BFR; This analysis compares the change over time in degrees of knee flexion between the BFR Therapy group and the No BFR Group from 2 weeks post-op to 12 weeks post-op. Underlying data was collected on a biweekly basis. This statistical test utilized the null hypothesis that there would be no difference between groups in the change in degrees of knee flexion over time; Test type: Equivalence — The a priori threshold for statistical significance was set at 0.05; p = 0.242, t-test, 1 sided

6. Primary Outcome: Degrees of Knee Extension
Description: Degrees of knee extension will be measured on the operative side by a licensed physical therapist, with zero degrees indicating the knee completely at extension and negative degrees indicating degrees of hyperextension. The outcome will be reported biweekly and then finally reported as a change in degrees from the first measurement to the final measurement. The results reported in this data table refer to the degrees of knee extension at each reported time point. The change in knee extension results can be found in the statistical analysis section.
Time Frame: Tracked in the perioperative week and then from initiation of therapy 2 weeks post-op through 12 weeks post-op.
Measure: Mean (Standard Error); unit: degrees
Arm/Group | BFR Therapy | No BFR
Number analyzed (Participants) | 25 | 20
degrees
  Perioperative week | -6.88 (1.40) | -5.25 (1.25)
  2 weeks post-op | -3.60 (1.45) | -3.20 (0.84)
  4 weeks post-op | -0.32 (0.73) | -0.09 (0.89)
  6 weeks post-op | 0.68 (0.51) | -0.15 (0.58)
  8 weeks post-op | 1.22 (0.64) | 0.63 (0.73)
  10 weeks post-op | 1.62 (0.68) | 0.33 (0.67)
  12 weeks post-op | 1.59 (0.63) | 0.31 (0.60)
Statistical Analysis 1: Comparison: BFR Therapy vs No BFR; This analysis compares the change over time in degrees of knee extension between the BFR Therapy group and the No BFR Group from 2 weeks post-op to 12 weeks post-op. Underlying data was collected on a biweekly basis. This statistical test utilized the null hypothesis that there would be no difference between groups in the change in degrees of knee extension over time; Test type: Equivalence — The a priori threshold for statistical significance was set at 0.05; p = 0.049, t-test, 1 sided

7. Secondary Outcome: Adverse Effects
Description: Observation of any adverse events associated with BFR therapy, such as numbness, cuff-site pain, and bruising.
Time Frame: Tracked from initiation of therapy 2 weeks post-op through 12 weeks post-op
Measure: Number; unit: adverse events
Arm/Group | BFR Therapy | No BFR
Number analyzed (Participants) | 25 | 20
adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | BFR Therapy | No BFR
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/20
Other Adverse Events (participants affected / at risk) | 0/25 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT03758755/Prot_SAP_000.pdf